CLINICAL TRIAL: NCT01578759
Title: Effects of Salpingectomy During Laparoscopic Hysterectomy on Ovarian Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-0440
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2014-10

CONDITIONS: Laparoscopic Hysterectomy
Keywords: ovarian function tests
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salpingectomy group (Experimental): Participants in this group will have their fallopian tubes removed.
  Interventions: Procedure: Salpingectomy
- No Salpingectomy Group (No Intervention): Participants in this group will not have their fallopian tubes removed.

INTERVENTIONS:
Procedure: Salpingectomy — Removal of the fallopian tubes
  Arms: Salpingectomy group

SUMMARY:
The purpose of this study is to assess the feasibility of performing a randomized clinical trial evaluating the effect of salpingectomy (removal of the fallopian tubes) during laparoscopic hysterectomy on ovarian function. The hypothesis is that removal of the tubes can prevent diseases of the fallopian tubes such as infection, hydrosalpinx (fluid-filled tubes)and additional invasive procedures such as further imaging work-ups and further surgery related to the tubes.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45 scheduled for laparoscopic hysterectomy with planned preservation of both ovaries.

Exclusion Criteria:

* Carrier for the gene that codes for breast cancer type 1 susceptibility protein (BRCA1) or the gene that codes for breast cancer type 2 susceptibility protein (BRCA 2).
* Personal history of gynecologic cancer
* Pregnancy
* Non-English speaking
* Unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ovarian function as measured by Anti-Mullerian Hormone (AMH) | AMH blood samples collected prior to surgery at day 1 (the day of the surgery) and at 1 and 3 months after day 1.

SECONDARY OUTCOMES:
Patient demographics | Prior to surgery
  The following routinely collected information will be included in the data analysis: age, body mass index, and surgery indication.
Patient surgical outcomes | Postoperatively on day 1
  The following surgical outcomes will be collected postoperatively: total operating time, estimated blood loss, surgical complications, and surgical pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Findley, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Division of Advanced Laparoscopy and Pelvic Pain, Department of Obstetrics and Gynecology, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Findley AD, Siedhoff MT, Hobbs KA, Steege JF, Carey ET, McCall CA, Steiner AZ. Short-term effects of salpingectomy during laparoscopic hysterectomy on ovarian reserve: a pilot randomized controlled trial. Fertil Steril. 2013 Dec;100(6):1704-8. doi: 10.1016/j.fertnstert.2013.07.1997. Epub 2013 Aug 29. PMID 23993887